CLINICAL TRIAL: NCT05031598
Title: Long-term Fasting: Multi-system Adaptations in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buchinger Wilhelmi Development & Holding GmbH (Other)
Collaborators: Buchinger Wilhelmi Clinic (Unknown); Claude Bernard University (Other); University of Milan (Other); Omegametrix GmbH (Unknown); King's College London (Other); MVZ Humangenetik Ulm (Unknown); University of Graz (Other); Leiden University Medical Center (Other); MVZ Labor Ravensburg (Unknown); ETH Zurich (Other)
Responsible Party: Principal Investigator, Françoise Wilhelmi de Toledo, Scientific Director; Principal Investigator, Buchinger Wilhelmi Development & Holding GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F-2021-075
Record Dates: First submitted 2021-08-11; First posted 2021-09-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Fasting
Keywords: long-term fasting; Buchinger Wilhelmi program; magnetic resonance imaging (MRI); magnetic resonance spectroscopy (MRS); HDL efflux capacity; fatty acid profile in erythrocyte membrane; gut microbiota; metabolomics; hydrogen sulfide and transsulfuration pathway
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: single-arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-term fasting (Experimental): The participants will undergo 6-12 fasting days according to the Buchinger Wilhelmi fasting program
  Interventions: Other: Long-term fasting according to the Buchinger Wilhelmi fasting program

INTERVENTIONS:
Other: Long-term fasting according to the Buchinger Wilhelmi fasting program — the participants will undergo a fasting program that includes the daily intake of 250 kcal under medical supervision

SUMMARY:
The aim of this trial is to investigate the effects of long-term fasting on size, mass, composition and function of metabolic active tissues in several organs that reexpand possibly rejuvenated after 1-4 months. Additionally, the lipid metabolism is investigated in depth.

DETAILED DESCRIPTION:
Fasting displays numerous positive effects on metabolism, health and aging. Surprisingly, few considerations are given to long-term fasting periods.

The metabolic switch from food-derived glucose to adipose tissue-derived fatty acids and ketones as primary cellular fuel is the key to fasting metabolism. Fasting has been shown to improve cardiovascular risk factors and gut microbiota in humans. It provokes profound changes in lipid metabolism. However, many questions are still open concerning the mobilization, exchange, and function of lipids during long-term fasting. Furthermore, recent results show the ability of periodic restrictive nutritional strategies to trigger organ regeneration. This promising regenerative power has not been investigated comprehensively in humans. In addition, the knowledge about the role of human faecal microbiota in health and disease is increasing. Only little is known about its composition and function during fasting. We found indications that the gut microbiome could influence energy metabolism and consequently could influence the dynamic of the metabolic switch.

Long-term fasting under medical supervision according to the Buchinger Wilhelmi fasting program has been demonstrated to be safe and well-tolerated.

The current project investigates the effects of a 9±3 days fasting period by a multi-systemic approach focusing on lipid metabolism and the gut microbiome in 100 subjects. Additionally, the body composition in combination with muscle performance will be analyzed in-depth in a subgroup of 32 subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 22 - 35 kg/m2

Exclusion Criteria:

* intake of medication (cardiovascular diseases, lipid and glucose metabolism)
* chronic manifest psychical and psychiatric diseases
* participation in another study
* pregnancy or breastfeeding
* in the MRI/MRS sub-study, any MRI contraindication (claustrophobia, pacemakers, MR-incompatible prosthetic valves, metallic implants, foreign metallic body)
* active uncontrolled gastrointestinal disorders including ulcerative colitis, Crohn's disease, indeterminate colitis, severe irritable bowel syndrome, persistent infectious gastroenteritis, persistent or chronic diarrhea of unknown etiology, recurrent Clostridium difficile infection
* major surgery of the GI tract, in the past five years. Any major bowel resection at any time
* intake of antibiotics in the last 2 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in whole body composition | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in the composition of the heart | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in the composition of the liver | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in the composition of the kidney | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in the composition of the spleen | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in the composition of the quadriceps | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in the composition of the adipose tissue | Baseline and changes at the end of fasting as well as one and four months afterwards
  Fat mass, lean mass, water content measured by magnetic resonance imaging
Changes in HDL cholesterol efflux capacity | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured in serum by a standardized used radioisotopic technique
Changes in serum cholesterol loading capacity | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured in serum using radioactive cholesterol loaded macrophages
Changes in HS-Omega-3 Index | Baseline and changes at the end of fasting as well as one and four months afterwards
  Determination of fatty acid (C 14:0; 16:0; 18:0; 20:0; 22:0; 24:0; 16:1 n-7; 18:1 n-9; 20:1 n-9; 24:1 n-9; 18:2 n-6; 18: 3 n-6; 20: 3 n-6; 22:2 n-6; 20:4 n-6; 22:4 n-6; 22:5 n-6; 18: 3 n-3; 20:5 n-3; 22:5 n-3; 22:6 n-3; 16:1 n-7t; 18:1 n-9t; 18:2 n-6tt; 18:2 n-6ct; 18:2 n-6tc) in erythrocyte membranes with highly standardized analytical procedure
Changes in faecal microbiota composition and function (carbohydrate metabolism) | Baseline and changes after an average of 10 (+/-3) fasting days
  Shotgun metagenomics, 5Gb of DNA sequencing data.
Changes in metabolome | Baseline and changes after 3 fasting days, the end of fasting as well as one and four months afterwards
  using an untargeted metabolomics approach to investigate changes in the metabolome, with a focus on the polyamine biosynthetic pathway at the cellular level in PBMCs and compare them with changes in the circulating plasma/serum metabolome
Changes in hydrogen sulfide production capacity | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured in serum and urine using the lead acetate assay

SECONDARY OUTCOMES:
Changes in brain morphometry | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured by magnetic resonance imaging
Changes in cardiac mass | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured by magnetic resonance imaging
Changes in lower limbs (quadriceps, hamstrings, calves) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured by magnetic resonance imaging
Changes in lumbosacral muscle mass | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured by magnetic resonance imaging
Changes in systolic cardiac function | Baseline and changes at the end of fasting as well as one and four months afterwards
  global and regional function (right and left ejection fraction, right and left end-diastolic and end-systolic volumes, peak regional strains (circumferential, longitudinal strain) measured with magnetic resonance imaging
Changes in diastolic cardiac function | Baseline and changes at the end of fasting as well as one and four months afterwards
  global and regional diastolic function (peak filling rate, torsion rate, diastolic strain rate) measured with magnetic resonance imaging
Changes in apparent diffusion coefficient (ADC) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with magnetic impedance imaging
Changes in fiber strain (Eff) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with magnetic impedance imaging
Changes in fractional anisotropy (FA) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with magnetic impedance imaging
Changes in helix angle (HA) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with magnetic impedance imaging
Changes in mean diffusivity (MD) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with magnetic impedance imaging
Changes in cardiovascular fitness | Baseline and changes at the end of fasting as well as one and four months afterwards
  using the maximal oxygen consumption (VO2max)
Changes in muscle metabolism and mitochondrial oxidative capacity: TauPCr(s) | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: PCr hydrolysis (%) | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: PCr concentration | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: Pi concentration | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: ATP concentration | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: pH at rest and post exercise in mM | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: T1 of metabolites at rest | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in muscle metabolism and mitochondrial oxidative capacity: PCr consumption | Baseline and changes at the end of fasting as well as one and four months afterwards
  during ergometric effort in MRI at the level of the sural muscle (31P spectroscopy)
Changes in multiparametric muscle quantification: T2 | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with quantitative magnetic impedance imaging
Changes in multiparametric muscle quantification: T2 * relaxation time | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with quantitative magnetic impedance imaging
Changes in multiparametric muscle quantification: susceptibility (chi) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with quantitative magnetic impedance imaging
Changes in multiparametric muscle quantification: fat fraction (PDFF) | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with quantitative magnetic impedance imaging
Changes in quadricipital maximum voluntary contraction | Baseline and changes at the end of fasting as well as one and four months afterwards
  measured with magnetic impedance imaging
Changes in DNA methylation | Baseline and changes at the end of fasting as well as one and four months afterwards
  biomarker of biological aging using erythrocytes
Changes in serum amyloid A levels | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum
Changes in paraoxonase (PON-1) activity | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum
Changes in lipoprotein transfer enzymes | Baseline and changes at the end of fasting as well as one and four months afterwards
  CETP activity, determined as U/ml using a commercially available assay
Changes in GlycA | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum
Changes in proprotein convertase subtilisin/kexin type 9 (PCSK9) | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum by ELISA
Changes in chylomicrons | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum
Changes in oxidized phospholipids | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum
Changes in enzymes | Baseline and changes after 3 fasting days, the end of fasting as well as one and four months afterwards
  immunoblotting of relevantly altered enzymes in PBMCs
Changes in persulfidation | Baseline, and changes after 3 fasting days, at the end of fasting as well as one and four months afterwards
  persulfidation in serum and urine
Changes in sulfur compounds | Baseline and changes after 3 fasting days, at the end of fasting as well as one and four months afterwards
  amino acids (using a targeted approach), thiosulfate (measured using the monobromobimane method using HPLC and LC-MS/MS), cysteine and cystine (use the S-sulfocysteine (SSC) method which is a HPLC-based method using automated precolumn derivatization with OPA and UV detection at 338 nm) in serum and urine
Changes in thiosulfate levels | Baseline and changes after 3 fasting days, at the end of fasting as well as one and four months afterwards
  measured using the monobromobimane method using HPLC and LC-MS/MS
Changes in cysteine and cystine levels | Baseline and changes after 3 fasting days, at the end of fasting as well as one and four months afterwards
  using the S-sulfocysteine (SSC) method which is a HPLC-based method using automated precolumn derivatization with OPA and UV detection at 338 nm in serum and urine
Changes in amino acids | Baseline and changes after 3 fasting days, at the end of fasting as well as one and four months afterwards
  using a targeted approach in serum and urine

OTHER OUTCOMES:
Changes in body weight | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  in kg
Changes in body mass index | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  in kg/m²
Changes in abdominal circumference | Baseline and changes at the end of fasting as well as one and four months afterwards
  in cm
Changes in resting systolic blood pressure | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  in mmHg
Changes in resting diastolic blood pressure | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  in mmHg
Changes in resting heart frequency | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  in beats/min
Changes in bio-electrical multifrequency impedance analysis | Baseline and changes at the end of fasting as well as one and four months afterwards
  Global and segmental body composition (water, fat and lean mass), liquid distribution (total, extracellular and intracellular water), metabolic indexes (metabolic activity index (MAI), protein content (total and active cell mass fraction) as determined by bioimpedance analysis
Changes in liver stiffness | Baseline, during and after fasting
  measured by FibroScan
Changes in physical activity | Before, daily during fasting as well as one and four months afterwards
  intensity, duration, frequency measured by triaxial actigraphy
Changes in circadian rhythm and sleep | Before, daily during fasting as well as one and four months afterwards
  measured by triaxial actigraphy
Changes in mental well-being | Baseline and at the end of fasting as well as one and four months afterwards
  questionnaires: Warwick-Edinburgh Mental Well-Being Scale
Changes in global health | Baseline and at the end of fasting as well as one and four months afterwards
  questionnaires: PROMIS Scale
Changes in physical activity | Baseline and at the end of fasting as well as one and four months afterwards
  questionnaires: Godin Leisure-Time Exercise Questionnaire
Changes in sleep quality | Baseline and at the end of fasting as well as one and four months afterwards
  questionnaires: Pittsburgh Sleep Quality Index
Changes in ketonuria | during the fasting period and food reintroduction
  Ketone bodies in urine measured by urine dip sticks
Changes in ketonemia | during the fasting period and food reintroduction
  Ketone bodies in capillary blood
Changes in glycemia | during the fasting period and food reintroduction
  Glucose in capillary blood
Changes in dietary behaviour | Baseline and after fasting as well as one and four months afterwards
  questionnaire: short healthy eating index survey
Changes in smoking behaviour | Baseline and after fasting as well as one and four months afterwards
  questionnaire
Changes in alcohol consumption | Baseline and after fasting as well as one and four months afterwards
  questionnaire
Changes in physical activity | Baseline and after fasting as well as one and four months afterwards
  in hours/week
Changes in energy level | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in emotional well-being | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in physical well-being | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: fatigue | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: muscle weakness | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: back pain | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: hunger | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: anxiety | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: headache | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Changes in symptoms: sleep disturbances | Baseline, daily during fasting and food reintroduction as well as one and four months afterwards
  measured by visual scale (0-10)
Adverse events | through study completion, an average of 4.5 months
  Documentation of side effects
Changes in blood count | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: leucocytes, erythrocytes, haemoglobin, haematocrit, MCV, MCH, MCHC, thrombocytes, bilirubin
Changes in differential blood count | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: basophiles, neutrophils, eosinophiles, monocytes, reticulocytes
Changes in coagulation | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: INR, PTT in sec
Changes in liver enzymes | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: GOT, GPT, GGT, AP in U/l
Changes in kidney parameters | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: uric acid, urea, creatinine in mg/dl
Changes in inflammatory parameters | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: hs-CRP, ESR in mm/h, inflammasome, cortisol in µg/dl
Changes in glucose metabolism | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: glucose in mmol/l, HbA1c in %, insulin in mU/l
Changes in lipid parameters | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: total cholesterol, HDL-C, LDL-C, triglycerides in mmol/l
Changes in electrolytes | Baseline and at the end of fasting as well as one and four months afterwards
  blood parameters: sodium, potassium, calcium, magnesium in mmol/l
Changes in the immune response to fasting | Baseline, after 3 fasting days, and at the end of fasting as well as one and four months afterwards
  using single cell nucleus sequencing
Changes in cell populations (natural killer and T cells) | Baseline, after 3 fasting days, and at the end of fasting as well as one and four months afterwards
  using single cell nucleus sequencing
Changes in lipoprotein subclasses | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum by high-density ultracentrifugation reflecting cholesterol and triglyceride composition
Changes in apolipoproteins | Baseline and changes at the end of fasting as well as one and four months afterwards
  ApoA-I and ApoB determined in serum
Changes in lipoprotein(a) | Baseline and changes at the end of fasting as well as one and four months afterwards
  determined in serum
Changes in methylation based clocks | Baseline and changes at the end of fasting as well as one and four months afterwards
  biomarker of biological aging using PBMCs
Sociodemographic Measurements | Baseline
  Age, gender, language, complete family history, current and previous illness and co-morbidities, and current medications
Changes in nitrogen balance | Baseline, daily during fasting as well as food reintroduction
  nitrogen in 24-hours-urine

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Wilhelmi de Toledo, Dr, Principal Investigator — Buchinger Wilhelmi Clinic
Locations (1):
- Buchinger Wilhelmi clinic, Überlingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grundler F, Palumbo M, Adorni MP, Zimetti F, Papotti B, Plonne D, Holley A, Mesnage R, Ruscica M, Wilhelmi de Toledo F. HDL cholesterol efflux capacity and cholesterol loading capacity in long-term fasting: Evidence from a prospective, single-arm interventional study in healthy individuals. Atherosclerosis. 2024 Oct;397:118548. doi: 10.1016/j.atherosclerosis.2024.118548. Epub 2024 Aug 6. PMID 39180960
- [Derived] Grundler F, Viallon M, Mesnage R, Ruscica M, von Schacky C, Madeo F, Hofer SJ, Mitchell SJ, Croisille P, Wilhelmi de Toledo F. Long-term fasting: Multi-system adaptations in humans (GENESIS) study-A single-arm interventional trial. Front Nutr. 2022 Nov 17;9:951000. doi: 10.3389/fnut.2022.951000. eCollection 2022. PMID 36466423